CLINICAL TRIAL: NCT06822075
Title: SANTE - Solidarité, Activités Sportives et Ludiques, Nouveauté, Tissu et Étudiants
Brief Title: Impact of a Physical Activity Program on the Mental Health of Medical Students.
Acronym: SANTE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: SANTE
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Health Behavior; Health Related Physical Fitness; Mental Health; Sedentary Behaviors; Physical Inactivity; Medical Student
Keywords: Health; Student; Curriculum; Behavior; Medical; Physical activity; Sedentary; Mental and physical health; Isolation; Loneliness
MeSH Terms: conditions — Health Behavior; Psychological Well-Being; Sedentary Behavior; Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: An interventional study (intervention = SANTE program) with a crossover protocol, preceded by an randomization (1:1). One group will get SANTE Program during the first period of the study, then noting during the second period.
  The other group will get noting during the first period of the study, then SANTE program during the second period. Both groups will successively benefit from the intervention (INT-1 group first, followed by the INT-2 group).
Who Masked: Participant
Masking Description: Participants will not know whether they are receiving the intervention first or second.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INT-1 (Experimental): The group INT-1 will get SANTE Program during the first period of the study, then noting during the second period.
  Interventions: Behavioral: SANTE program
- INT-2 (Experimental): The group INT-2 will get noting during the first period of the study, then SANTE program during the second period.
  Interventions: Behavioral: SANTE program

INTERVENTIONS:
Behavioral: SANTE program — The intervention will consist of distinct period. Fisrt, 3 complete assessment periods will be realized : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16) for evaluate the evolution of the health-related behavior, mental and physical health. Second, the SANTE program intervention will be implemented. Intervention 1 (week 3 and 7) for INT-1 group receive the SANTE program and INT-2 group do noting ; Intervention 2 (week 10-14) for INT-2 group receive the SANTE program and INT-1 do noting.
  The SANTE intervention will consist of (at a minimum):
  * 1 to 2 group physical activity sessions per week
  * 1 outdoor outing (full-day or half-day) per month
  * 1 individual meeting with a physical activity and sports expert

SUMMARY:
University students frequently adopt a sedentary lifestyle with low levels of physical activity, leading to a deterioration in their health. A significant number of them also suffer from social isolation. Moreover, numerous studies have highlighted the vulnerability of university students (particularly those in medical programs) to mental health issues. Medical students, with their demanding academic curriculum, are no exception to this trend.

A student association at the Lyon Est Faculty of Medicine reported that students' mental health is very low (2022): at least 1 in 2 students has experienced a depressive episode, and 1 in 3 has had suicidal thoughts during their studies. Other recent studies indicate that medical students at Lyon Est exhibit high levels of stress, low self-confidence, and excessive sedentary behavior (ECOSTRESS and ECOSPERF studies, 2021, 2022, and 2023). Unfortunately, in 2024, new mental health surveys among medical students from the second year through the end of their internship continue to confirm these findings.

The SANTE project aims to offer solution to student to a highly effective means of improving both their mental health and their level of physical activity throught an intervention program. More precisely, the goal of this interventional study is to evaluate the impact of a physical activity program on the mental health in second-cycle medical students at the University of Lyon 1. The development of the SANTÉ program was based on (i) data from the literature, (ii) results from a previous local study (IRB No. 2024-07-02-03) that identified student needs through individual interviews and focus groups, and (iii) local findings from a co-construction workshop with students.

ELIGIBILITY:
Inclusion Criteria:

* Being a 2th-year or a 3th-year medical student at the Faculty of Medicine Lyon East and Lyon South during the academic years 2024-2025.
* Having read the information note.
* Having signed the written consent.

Exclusion Criteria:

* No exclusion criteria will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall mental health : Evolution of the score obtained at the Depression Anxiety and Stress Scale-21 (DASS-21) | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of overall mental health will be assessed through the DASS-21 questionnaire. A total score can also be assessed ranging from 0 (normal) to 63 (extremely severe). A score for the three subscales (depression, anxiety, stress) can also be assessed, each score ranging from 0 (normal) to 21 (extremely severe).
  The measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).

SECONDARY OUTCOMES:
Perceived level of physical activity : Score obtained at the Onaps-PAQ on physical activity levels. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of physical activity and sedentary will be assessed through the Onaps-PAQ (National Observatory for Physical Activity and Sedentariness - Physical Activity Questionnaires) during a typical week. Scores are expressed in hours per day for week and weekend days. This measure will be done during the 3 complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Perceived level of well-being : Score obtained at The World Health Organization-Five (WHO-5) Well-Being Index | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of well-being will be assessed through the WHO-5 WELL-BEING index. The total score is ranging from zero (worst possible mental well-being) to 100 (best possible mental well-being).
  This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Perceived level of stress : Score obtained at the Perceveid Stress Scale (PSS) | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The student's level of stress will be assessed through the PSS questionnaire ranging from 0 (none) to 40 (extreme).This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Perceived level of loneliness : Score obtained at the UCLA Loneliness Scale. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of loneliness will be assessed through the UCLA Loneliness Scale ranging from 20 (low) to 80 (extreme). This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Perceived level of sleep disturbance : Score obtained at the Pittsburgh Sleep Quality Index (PSQI) | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of sleep disturbance will be assessed through the Pittsburgh Sleep Quality Index (PSQI) ranging from 0 (none) to 21 (extreme). This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Perceived level of fatigue : Score obtained at the Multidimentional Fatigue Inventory (MFI) | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The student's level of fatigue will be assessed through the MFI questionnaire that covers various dimensions of fatigue, including general fatigue (9 to 45), mental fatigue (6 to 30), reduced motivation (2 to 10), and reduced activity (3 to 15). The higher the score, the greater the fatigue. This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Habits and beliefs about physical activity : Scores obtained at the Habits and Beliefs About Physical Activity Questionnaire | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  Participants' habits and beliefs about physical activity will be assessed through this 9-item questionnaire, with responses ranging from 1 (strongly agree) to 5 (strongly disagree). This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Physical Fitness markers - Strength. The force developed during a maximal isometric contraction of the quadriceps. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students basal level of physical fitness will be assessed through a muscular strength test. This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Physical Fitness markers markers - Power. Height of jump. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students basal level of physical fitness will be assessed through a power test, a vertical jump. The squat jump is plyometric exercise in which a person bends their knees to lower their body into a squat position, then performs an explosive jump upwards by extending the hips, knees, and ankles simultaneously. During this exercise, the height of jump will be measured.This measure will be done during the 3 complete complete assessment periods : pre-intervention (week 1-2) ; mid-intervention (week 8-9) ; post-intervention (week 15 - 16).
Physical Fitness markers markers - Power. Height of jump. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of physical fitness will be assessed through a power test, a vertical jump. The squat jump is plyometric exercise in which a person bends their knees to lower their body into a squat position, then performs an explosive jump upwards by extending the hips, knees, and ankles simultaneously. During this exercise, the height of jump will be measured.
Physical Fitness markers - Endurance. Speed through the endurance test. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of physical fitness will be assessed through cardiorespiratory endurance test (modified VAMEVAL). During this test, the velocity at maximal aerobic (VMA) is the maximum speed (velocity) reached where the individual can still maintain aerobic metabolism without transitioning into anaerobic metabolism. VO2max refers to the maximum rate of oxygen consumption during intense exercise, typically measured in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). It is a key indicator of an individual's cardiovascular fitness and aerobic endurance.
Physical Fitness markers - Endurance. Heart rate during the endurance test. | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of physical fitness will be assessed through a cardiorespiratory endurance test (modified VAMEVAL). The heart rate will be measured at three moments: maximum, submaximal, at 1 minute, and 3 minutes of recovery.
Physical Fitness markers - Flexibility. Lower body | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of flexibility of lower body will be assessed through the sit and reach test.
Physical Fitness markers - Flexibility. Upper body | Week 1 and 2 (pre-intervention) Week 8-9 (mid-intervention) Week 15-16 (Post-intervention)
  The students level of flexibility will be assessed through a upper body test.

OTHER OUTCOMES:
Likert - Questionnaire of satisfaction | Week 15-16 (Post-intervention)
  The perceived level of the satisfaction ("Are you satisfied with the intervention ?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 4 (very satisfied). The measure will be done during the post-intervention (week 15 - 16).

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schlatter, Dr., Principal Investigator — RESHAPE U1290 INSERM UCBL-LYON 1 Rockfeller, Lyon France.
Locations (1):
- RESHAPE, Lyon, France, France

IPD SHARING:
Plan to Share IPD: Undecided